CLINICAL TRIAL: NCT04039048
Title: Effects of Cerebellar Transcranial Direct Current Stimulation During Balance Training on Cerebellar Ataxia
Brief Title: Effect of ctDCS During Balance Training on Cerebellar Ataxia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Study director, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: cerebellarataxia_balance_ctDCS
Record Dates: First submitted 2019-07-28; First posted 2019-07-31 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Cerebellar Ataxia; Cerebellum; Injury; Balance
Keywords: Biodex balance system; Posture control; Ataxia' severity; ctDCS
MeSH Terms: conditions — Cerebellar Ataxia; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ctDCS during Balance training (Experimental)
  Interventions: Device: cerebellar transcranial direct current stimulation; Other: Balance training
- ctDCS sham during Balance training (Sham Comparator)
  Interventions: Device: Sham cerebellar transcranial direct current stimulation; Other: Balance training

INTERVENTIONS:
Device: cerebellar transcranial direct current stimulation — Non-invasive brain stimulation technique is able to modulate the brain activity through a low-intensity current. The anodal will be positioned 1 cm below inion and cathodal in the right deltoid muscle. 20 minutes with a 2mA current.
  Other Names: ctDCS
  Arms: ctDCS during Balance training
Device: Sham cerebellar transcranial direct current stimulation — Non-invasive brain stimulation technique is able to modulate the brain activity through a low-intensity current. The anodal will be positioned 1 cm below inion and cathodal in the right deltoid muscle. 30 seconds with a 2mA current.
  Other Names: ctDCS sham
  Arms: ctDCS sham during Balance training
Other: Balance training — Balance training will be performed through the Biodex Balance System for 20 minutes.

SUMMARY:
Cerebellar ataxia is a neurologic symptom caused by damage or dysfunction in the cerebellum and its pathways that results in loss of coordination, balance and postural control. There is a high rate (93%) of fallings for this population that could limit daily life activities. Pharmacological interventions are not able to modify the balance, therefore, new approaches to rehabilitate must be studied. ctDCS is a non-invasive brain stimulation that seems to be a new and innovator technique to restore ataxia symptoms. The purpose of this study is to evaluate the effects of ctDCS associated with balance training on cerebellar ataxia patients. A counterbalanced crossover, sham-controlled, triple blind trial will be performed. All subjects will receive the real and sham ctDCS associated to balance training. The anodal ctDCS (2 mA, 20 minutes) or sham (2mA, 30 seconds) will be applied during balance training at Biodex Balance System (BBS). The balance will be the primary outcome and will be evaluated through Posture Control at Biodex Balance System. Ataxia' severity and functional mobility will be the secondary outcomes and will be evaluated by the scale for the assessment and rating of ataxia (SARA) and 10 meters walking test, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Cerebellar ataxia
* Score > 1 ≤ 4 on posture of Scale for assessment and rating of ataxia

Exclusion Criteria:

* Individuals with other neurological disorders, postural hypotension, vestibular, visual, cardiovascular or musculoskeletal disorders that affect the performance of the proposed tests;
* Pacemaker;
* History of seizures;
* Metallic implants in the head or neck;
* Medication change (3 months) during the period of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Change in balance | 5 minutes before the intervention and 10 minutes after the intervention
  The change in balance will be assessed through postural control index of Biodex Balance System. This postural control index is a continuous variable where lower index means less instability and better balance.

SECONDARY OUTCOMES:
Change in Ataxia' severity | 10 minutes before the intervention and 15 minutes after the intervention
  The ataxia' severity will be assessed by the Scale for the Assessment and Rating of Ataxia (SARA). It consists of eight items (gait, stance, sitting, speech disturbance, finger chase, nose-finger test, fast alternating, hand movements, and heel-shin slide), where higher score (40) mean more severe ataxia, whereas lower score (0) means less ataxia symptoms. The score happens about the sum of the eight items.
Change in functional mobility | 15 minutes before the intervention and 20 minutes after the intervention
  The patient will walk 10 meters and the time will be measured to determine the functional mobility. Where lower time to walk 10 meters, better functional mobility.

CONTACTS AND LOCATIONS:
Locations (1):
- Kátia Monte-Silva, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Brito R, Fabricio JV, Araujo A, Barreto G, Baltar A, Monte-Silva K. Single-Session Cerebellar Transcranial Direct Current Stimulation Improves Postural Stability and Reduces Ataxia Symptoms in Spinocerebellar Ataxia. Cerebellum. 2024 Oct;23(5):1993-2002. doi: 10.1007/s12311-024-01696-9. Epub 2024 May 2. PMID 38693314